CLINICAL TRIAL: NCT07104851
Title: Efficacy and Sustainability of a Hybrid Psychological Intervention Integrating Resilience Theory and the Satir Model on Depression, Resilience, and Quality of Life in Adolescents: A Multi-center, Randomized Controlled Trial
Brief Title: A Hybrid Psychological Intervention for Depression in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kenan Ren, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-S00443
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Resilience-Satir Hybrid Intervention Group (Experimental): In addition to treatment as usual (TAU), participants received a structured 12-week group nursing intervention program. The program consisted of one 90-minute session per week, co-facilitated by trained psychiatric nurses. The intervention included three modules: Module 1 (Weeks 1-4) focused on safety and identifying emotions using Satir's "Iceberg" metaphor and personal strengths; Module 2 (Weeks 5-8) focused on building skills in problem-solving, cognitive reframing, and congruent communication; Module 3 (Weeks 9-12) focused on integrating skills and future-planning.
  Interventions: Behavioral: Resilience-Satir Hybrid Intervention
- Active Comparator: Treatment as Usual (TAU) Group (Active Comparator): Participants received standard care, which included regular psychiatric assessments, pharmacotherapy as deemed appropriate by the treating psychiatrist (primarily SSRIs), and routine nursing care. Routine care consisted of general health education, basic supportive communication, and monitoring of symptoms and side effects. No structured psychotherapy was provided.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Resilience-Satir Hybrid Intervention — A structured, 12-week, group-based psychological intervention integrating principles from Resilience Theory and the Satir Model to enhance coping skills, self-esteem, communication, and family dynamics.
  Arms: Experimental: Resilience-Satir Hybrid Intervention Group
Other: Treatment as Usual (TAU) — Standard care for adolescent depression, including pharmacotherapy and routine nursing support, without structured psychotherapy.
  Arms: Active Comparator: Treatment as Usual (TAU) Group

SUMMARY:
This multi-center, randomized controlled trial was conducted to evaluate the efficacy and long-term effects of a novel hybrid psychological intervention, which combines Resilience Theory with the Satir Model, for adolescents diagnosed with depression. The study compared this intervention to treatment as usual (TAU) to determine its impact on depressive symptoms, psychological resilience, self-esteem, and overall quality of life.

DETAILED DESCRIPTION:
Adolescent depression is a significant and growing public health concern. Traditional therapies have limitations, highlighting a need for innovative, engaging interventions. This study was designed to address this gap by developing and testing a hybrid model that integrates the strengths-based approach of Resilience Theory with the systemic, humanistic principles of the Satir Model. The study hypothesized that this combined intervention would be more effective than standard care in not only alleviating depressive symptoms but also in building lasting psychosocial resources. A total of 420 adolescents with depression were randomized to either the 12-week hybrid intervention group or a control group receiving treatment as usual. The intervention program was structured in three modules focusing on self-awareness, skill-building, and future-orientation. Outcomes were assessed at baseline, immediately post-intervention (12 weeks), and at a 6-month follow-up to evaluate the sustainability of the effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a major depressive episode according to DSM-5 criteria, confirmed by two independent psychiatrists.
* First episode, with a duration of 4 weeks to 12 months.
* Age between 13 and 18 years.
* HAMD-17 score ≥ 17.
* Capable of normal communication.
* Provision of informed consent by both the adolescent and legal guardians.

Exclusion Criteria:

* Lifetime diagnosis of bipolar disorder, schizophrenia, or other psychotic disorders.
* Depression secondary to a general medical condition or substance use.
* Acute suicidal risk (score ≥ 4 on MADRS item 10) requiring immediate intensive care.
* Currently receiving structured psychotherapy.
* Severe neurological or physical illness that could interfere with participation.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms as Measured by the 17-item Hamilton Depression Rating Scale (HAMD-17) | Baseline, 12 weeks, 6-month follow-up
  A clinician-rated scale assessing the severity of depression. Total scores range from 0 to 52. A lower score indicates a better outcome.
Change in Depressive Symptoms as Measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, 12 weeks, 6-month follow-up
  A clinician-rated scale sensitive to changes in core depressive symptoms. Total scores range from 0 to 60. A lower score indicates a better outcome.
Change in Depressive Symptoms as Measured by the Beck Depression Inventory-II (BDI-II) | Baseline, 12 weeks, 6-month follow-up
  A 21-item self-report questionnaire assessing the severity of depression. A lower score indicates a better outcome.

SECONDARY OUTCOMES:
Change in Psychological Resilience as Measured by the Resilience Scale for Chinese Adolescents (RSCA) | Baseline, 12 weeks, 6-month follow-up
  A 27-item self-report scale assessing personal strength and support strength. A higher score indicates better resilience.
Change in Self-Esteem as Measured by the Feelings of Inferiority Scale (FIS) | Baseline, 12 weeks, 6-month follow-up
  A 36-item self-report scale measuring self-esteem. A higher score indicates higher self-esteem and a better outcome.
Change in Coping Styles as Measured by the Simplified Coping Style Questionnaire (SCSQ) | Baseline, 12 weeks, 6-month follow-up
  A 20-item self-report measure assessing positive and negative coping styles. An increase in the positive coping subscale score indicates a better outcome.
Change in Medication Adherence as Measured by the Medication Adherence Rating Scale (MARS) | Baseline, 12 weeks, 6-month follow-up
  A 10-item self-report scale assessing medication compliance behavior and attitudes. A higher score indicates better adherence.
Change in Family Function as Measured by the Family APGAR Index | Baseline, 12 weeks, 6-month follow-up
  A 5-item screening tool to assess an individual's perception of family function (Adaptation, Partnership, Growth, Affection, Resolve). A higher score indicates better family function.
Change in Social Support as Measured by the Perceived Social Support Scale (PSSS) | Baseline, 12 weeks, 6-month follow-up
  A 12-item scale measuring perceived support from family, friends, and significant others. A higher score indicates better perceived social support.
Change in Quality of Life as Measured by the World Health Organization Quality of Life-BREF (WHOQOL-BREF) | Baseline, 12 weeks, 6-month follow-up
  A 26-item self-report a measure assessing quality of life across four domains: physical health, psychological health, social relationships, and environment. Higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China